CLINICAL TRIAL: NCT01813643
Title: A Multiple-Center, Randomized, Double-Blind Study of Comparison of Risperidone and Aripiprazole for Treatment
Brief Title: A Comparison of Risperidone and Aripiprazole for Treatment of Patirnts With Methamphetamine-Associated Psychosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Effects of aripiprazole was not obvious and showed adverse reaction obviously
Sponsor: Wei Hao (Other)
Responsible Party: Sponsor-Investigator, Wei Hao, The Second Xiangya Hospital of Cental South University, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100000-068941
Record Dates: First submitted 2012-08-19; First posted 2013-03-19 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine-Associated Psychosis; Aripiprazole; Risperidone
MeSH Terms: interventions — Risperidone; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Experimental): Aripiprazole arm,5mg/pill,20-30mg/day,non-forced titration method.last2-4weeks.
  Interventions: Drug: Aripiprazole
- Risperidone (Active Comparator): Risperidone arm and placebo tables,1mg/pill,2mg-6mg/day,non-forced titration method.last2-4weeks.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — Risperidone group,1mg/pill,2mg-6mg/day non-forced titration method,last 2-4weeks
  Other Names: Risperdal H20070057
  Arms: Risperidone
Drug: Aripiprazole — Aripiprazole group,5mg/pill,20mg-30mg/day non-forced titration method,last 2-4weeks
  Other Names: Aopai H20041507
  Arms: Aripiprazole

SUMMARY:
Methamphetamine-associated psychosis (MAP) has been considered a pharmacological or environmental pathogen model of schizophrenia (SCZ) due in part to similarities in clinical presentation (i.e. paranoia, hallucinations, disorganized speech, and negative symptoms), response to treatment (e.g.neuroleptics),and pathologic mechanisms (e.g. central dopaminergic neurotransmission) of both conditions. Both risperidone and aripiprazole are second generation antipsychotics，but have different pharmacological effects of antipsychotic treatment.This study was designed to examine the acute efficacy, safety, and tolerability of risperidone and aripiprazole for patients with MAP.

DETAILED DESCRIPTION:
Methods:A Multiple-Center, Randomized, Double-Blind.

ELIGIBILITY:
Inclusion Criteria:

1. Patients,Diagnostic and Statistical Manual of Mental Disorders 4thed. (DSM-IV) criteria for Methamphetamine-Associated Psychosis.
2. Must sign a Information consent form.
3. Required to provide detailed address and phone number

Exclusion Criteria:

1. Serious organic disease.
2. Suicide ideation or hurt others.
3. Taking antipsychotic within two weeks before.
4. drug allergy to Risperidone or Aripiprazole.
5. pregnancy and breastfeeding women.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The severity of psychosis | up to 4 weeks. participants will be followed for the duration of hospital stay
  Positive and Negative Syndrome Scale

SECONDARY OUTCOMES:
adverse drug reaction | up to 4 weeks. participants will be followed for the duration of hospital
  Barnes Scale , Simpson-Angus Scale , Abnormal Involuntary Movement Scale
Clinical general status | up to 4 weeks. participants will be followed for the duration of hospital stay
  Clinical general rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hao, MD., Ph.D., Study Director — Central South University
Locations (1):
- The Second Xiangya Hospital of Central University, Changsha, Hunan, China